CLINICAL TRIAL: NCT03190122
Title: Neurocognitive Outcome Assessment in Patients With Peri-optic Meningiomas After Excision With Or Without Pealing Of The Outer Layer Of The Cavernous Sinus: A Randomized Controlled Single Blinded Trial.
Brief Title: Neurocognitive Outcome Assesment in Patients With Peri-optic Meningiomas After Excision With Or Without Pealing Of The Outer Layer Of The Cavernous Sinus: A Randomized Controlled Single Blinded Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Hegazy, professor of neurosurgery, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-71-2016
Record Dates: First submitted 2017-05-10; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Neurocognitive Outcome Assesment in Patients With Perioptic Meningiomas

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with pealing of the outer layer of cavernous sinus (Active Comparator): Neurocognitive Outcome Assesment in Patients With Peri-optic Meningiomas After Excision With Pealing Of The Outer Layer Of The Cavernous Sinus
  Interventions: Procedure: surgical excision of the tumor
- group without pealing of the outer layer of cavernous sinus (Experimental): Neurocognitive Outcome Assesment in Patients With Peri-optic Meningiomas After Excision Without Pealing Of The Outer Layer Of The Cavernous Sinus
  Interventions: Procedure: surgical excision of the tumor

INTERVENTIONS:
Procedure: surgical excision of the tumor — Neurocognitive Outcome Assesment in Patients With Peri-optic Meningiomas After Excision With Or Without Pealing Of The Outer Layer Of The Cavernous Sinus: A Randomized Controlled Single Blinded Trial. [NCT ID not yet assigned]

SUMMARY:
Neurocognitive Outcome Assesment in Patients With Peri-optic Meningiomas After Excision With Or Without Pealing Of The Outer Layer Of The Cavernous Sinus: A Randomized Controlled Single Blinded Trial.

ELIGIBILITY:
Inclusion Criteria:

* preoptic meningioma, not recurrent, size is operative.

Exclusion Criteria:

* other meningiomas than preoptic , recurrent cases, size is not operative, other medical conditions affect the mental condition of the patient.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Outcome Assessment using MOCA scale | 1 year
  aggregated by our researchers in data base system in our department.

SECONDARY OUTCOMES:
Neurocognitive Outcome using neuropsychological assessment questionnaire | 1 year
  aggregated by our researchers in data base system in our department.